CLINICAL TRIAL: NCT00423072
Title: Middle Ear Pressure Disregulation in Cleft Palate Patients: Form-Function Correlates
Brief Title: Middle Ear Pressure Disregulation in Cleft Palate Patients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Cuneyt M. Alper, Professor, Otolaryngology, University of Pittsburgh
Other Study IDs: 0607009; 1P50DC007667 (NIH)
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Cleft Palate
Keywords: cleft palate; palatoplasty; otitis; middle ear; Eustachian tube
MeSH Terms: conditions — Cleft Palate; Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: children with cleft palate birth-24 months of age

SUMMARY:
The investigators know that middle-ear disease is very common in infants with cleft palate and causes hearing loss that can last into childhood. It is thought that a poor ability to keep the pressure in the middle ear at a similar level to that in the environment causes middle-ear disease and that this depends on the opening function of a natural tube that connects the back of the nose with the middle ear, called the Eustachian tube. The investigators believe that the middle-ear disease in cleft palate infants and children is caused by poor Eustachian tube function that in turn is caused by anatomical problems in the muscles that open the tube. The investigators plan to test these relationships by studying the changes between 5-24 months and 6 years in middle-ear health, the way the Eustachian tube works and Eustachian tube anatomy in cleft palate children.

DETAILED DESCRIPTION:
Otitis media with effusion (OME) is recognized as nearly universal in the population of infants and children with cleft palate (CP) and is often associated with long-standing conductive and, perhaps, sensorineural hearing losses. Most evidence suggests that OME in CP patients is a complication of inefficient Eustachian tube function (ETF). The investigators plan to use our most complete tests to characterize ETF in CP infants tested at age 5-24 months and followed up through age 6 years by yearly collection of clinical data for the presence/absence of OME and repeat ETF testing. To obtain anatomical data, the investigators will obtain basal and lateral cephalograms at age 3 years in all subjects and perform MRI tests prepalatoplasty when possible and then at 3 and 5 years on a subset of the enrolled children. Functional-anatomical reconstructions based on the MRI data will be studied for the mechanical interactions underlying the phenomenon of ET constriction in CP patients and examined for the possibility of surgical interventions to correct identified abnormal interactions.

ELIGIBILITY:
Inclusion Criteria:

* birth-24 months
* unrepaired or recently repaired cleft palate

Exclusion Criteria:

* cleft palate associated with syndrome
* known immune deficiency

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cleft palate <2 years of age
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2006-08; Primary Completion 2017-03-27 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
otitis media | 5 years
  status of middle ear at 5 years of age

SECONDARY OUTCOMES:
anatomic variables | 3 and 5 years
  MRI data at 3 and 5 years in subset; cephalometric x-rays at 6 yr.
Eustachian tube function testing | pre- and post palatoplasty, yearly to age 18 yrs
  either Forced Response testing or pressure chamber testing

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- ENT Research Center Childrens' Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alper CM, Losee JE, Mandel EM, Seroky JT, Swarts JD, Doyle WJ. Pre- and post-palatoplasty Eustachian tube function in infants with cleft palate. Int J Pediatr Otorhinolaryngol. 2012 Mar;76(3):388-91. doi: 10.1016/j.ijporl.2011.12.017. Epub 2012 Jan 9. PMID 22230559
- [Result] Alper CM, Losee JE, Mandel EM, Seroky JT, Swarts JD, Doyle WJ. Postpalatoplasty Eustachian tube function in young children with cleft palate. Cleft Palate Craniofac J. 2012 Jul;49(4):504-7. doi: 10.1597/11-065. Epub 2011 Jul 8. PMID 21740160
- [Result] Alper CM, Losee JE, Seroky JT, Mandel EM, Richert BC, Doyle WJ. Resolution of Otitis Media With Effusion in Children With Cleft Palate Followed Through Five Years of Age. Cleft Palate Craniofac J. 2016 Sep;53(5):607-13. doi: 10.1597/15-130. PMID 27533493